CLINICAL TRIAL: NCT04426292
Title: SARS-COV-2 Seroprevalence and Seroconversion Among Employees of the Universitair Ziekenhuis Brussel During the 2020 COVID-19 Outbreak
Acronym: COVEMUZ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: COVEMUZ
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-06

CONDITIONS: Sars-CoV2
MeSH Terms: interventions — COVID-19 Serological Testing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- General arm (Other): All patients follow this arm. Patients will undergo 3 blood sample testings at 3 different time points and have to fill in a questionnaire at 3 different time points
  Interventions: Diagnostic Test: Serological testing

INTERVENTIONS:
Diagnostic Test: Serological testing — Antibody testing for Sars-COV-2 antibodies in blood.

SUMMARY:
A novel zoonotic coronavirus was discovered in Wuhan (Hubei Province, China) mid-December 2019 and was named severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). The virus rapidly spread to the rest of the world, including Europe and explicitly affects the respiratory system, generating Coronavirus disease 2019 (COVID-19).

This study is a monocentric interventional prospective cohort study. After signing a written informed consent, participants will be recruited for questionnaire completion and blood sampling. Sample storage and analysis will be performed at the laboratory of microbiology of the UZ Brussel.

* To document SARS-CoV-2 seroprevalence among employees of the UZ Brussel at day 0 (i.e. at beginning of the study, planned early May 2020), month 2 and month 5.
* To document number of SARS-CoV-2 seroconversions among employees of the UZ Brussel over a period of 5 months.

ELIGIBILITY:
Inclusion Criteria:

* Any adult employee of the UZ Brussel who provided a signed informed consent to participate in the study.

Exclusion Criteria:

* UZ Brussel employees whose contract expires within 6 months of study initiation, with the exception of resident trainees (if training continues in another hospital, resident trainees will be asked to perform the last sampling when leaving the UZ Brussel).
* Staff not active during the inclusion period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2020-05-12 (Actual); Primary Completion 2021-12-23 (Estimated); Study Completion 2021-12-25 (Estimated)

PRIMARY OUTCOMES:
Seroprevalence | Change from baseline to 2 months and 5 months timepoint
  - To document SARS-CoV-2 seroprevalence among employees of the UZ Brussel at day 0 (i.e. at beginning of the study, planned early May 2020), month 2 and month 5.
seroconversions | Change from baseline to 2 months and 5 months timepoint
  - To document number of SARS-CoV-2 seroconversions among employees of the UZ Brussel over a period of 5 months.

SECONDARY OUTCOMES:
Incidence of definite cases | Change from baseline to 2 months and 5 months timepoint
  - To document the incidence of new definite cases of COVID-19 (based on self-reported positive PCR testing on nasopharyngeal swab) among employees of the UZ Brussel over a period of five months.
Incidence of probable cases | Change from baseline to 2 months and 5 months timepoint
  - To document the incidence of new probable cases of COVID-19 (based on study questionnaire) among employees of the UZ Brussel over a period of five months.
Antibody kinetics | Change from baseline to 2 months and 5 months timepoint
  - To document the SARS-CoV-2 antibody kinetics after confirmed and probable COVID-19. Specifically (1) electrostatic interactions, (2) dispersion forces, (3) hydrogen bonds, and (4) hydrophobic interactions.
Potential work-related risk factors | Change from baseline to 2 months and 5 months timepoint
  - To investigate potential work-related risk factors for SARS-CoV-2 infection among employees of the UZ Brussel.
Proportion of asymptomatic seroconversions | Change from baseline to 2 months and 5 months timepoint
  - To quantify the proportion of asymptomatic seroconversions among employees of the UZ Brussel over a period of five months.
Concerns for safety for infection with COVID-19 | Change from baseline to 2 months and 5 months timepoint
  - To document the concerns of HCW and non-HCW about their safety for infection with COVID-19.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided